CLINICAL TRIAL: NCT02220517
Title: A Prospective Randomized Study Comparing the Diagnostic Efficacy of MR-guided in Bore Prostate Biopsy Versus MRI/US Fusion-guided Prostate Biopsy in Men With at Least One Negative Prostate Biopsy
Brief Title: Randomized Study Comparing MR-guided in Bore Versus MRI/US Fusion-guided Prostate Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 003
Record Dates: First submitted 2014-07-07; First posted 2014-08-20 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Prostate Cancer
Keywords: MRI/US fusion-guided prostate biopsy; MR-guided in-bore prostate biopsy; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: MR-guided in-bore prostate biopsy (Experimental): Patients of arm A receive a targeted MR-guided in-bore prostate biopsy. From each prostate lesion defined in the diagnostic multiparametric MRI two targeted biopsy cores will be taken.
  Interventions: Device: MR-guided in-bore prostate biopsy
- B: MRI/US fusion-guided prostate biopsy (Experimental): Patients of arm B receive a targeted MRI/US fusion-guided prostate biopsy. From each prostate lesion defined in the diagnostic multiparametric MRI two targeted biopsy cores will be taken. Immediately after targeted biopsy patients undergo additional systematic TRUS-guided biopsy (12 biopsy cores)
  Interventions: Device: MRI/US fusion-guided prostate biopsy

INTERVENTIONS:
Device: MR-guided in-bore prostate biopsy — Patients of arm A receive a targeted MR-guided in-bore prostate biopsy. From each prostate lesion defined in the diagnostic multiparametric MRI two targeted biopsy cores will be taken.
  Arms: A: MR-guided in-bore prostate biopsy
Device: MRI/US fusion-guided prostate biopsy — Patients of arm B receive a targeted MRI/US fusion-guided prostate biopsy. From each prostate lesion defined in the diagnostic multiparametric MRI two targeted biopsy cores will be taken. Immediately after targeted biopsy patients undergo additional systematic TRUS-guided biopsy (12 biopsy cores)
  Arms: B: MRI/US fusion-guided prostate biopsy

SUMMARY:
The hypothesis of the study is that targeted MRI/US fusion-guided prostate biopsy with additional systematic transrectal ultrasound (TRUS)-guided biopsy significantly detects more prostate cancers than targeted MR-guided in-bore prostate.

DETAILED DESCRIPTION:
In men with previously negative prostate biopsy and persistent elevated prostate-specific antigen (PSA) value, it is unclear which strategy offers the highest detection rate for prostate cancer. The hypothesis of this study is that targeted MRI-guided biopsy combined with transrectal ultrasound (TRUS)-guided biopsy may potentially detect more cancers than MRI-guided prostate biopsies alone.

Men with at least one previously negative TRUS-guided biopsy and persistently elevated PSA values will be submitted to a multiparametric MRI examination of the prostate. Subsequently, all participants will be randomized (1:1) into both study arms. In study arm A patients will be submitted to targeted prostate biopsy based on the multiparametric MRI findings. Targeted biopsies will be performed using MRI-guided in-bore prostate biopsy. In study arm B targeted biopsies will be performed using MRI/TRUS-fusion-guided prostate biopsy with software-registration (MRI/TRUS image fusion). Patients of study arm B undergo additional systematic 12-core TRUS-guided prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

* At least one prior negative prostate biopsy
* Prostate-specific antigen (PSA) > 4 ng/ml

Exclusion Criteria:

* Known prostate cancer
* Contraindications against MRI
* Contraindications against prostate biopsy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2011-11; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Prostate cancer detection rate | 1 week after biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Christian Arsov, MD, Principal Investigator — Department of Urology, University of Düsseldorf
Locations (1):
- University Hospital Düsseldorf, Düsseldorf, Germany